CLINICAL TRIAL: NCT02904772
Title: An Open Label, Multi-centre Trial of Alipogene Tiparvovec for the Treatment of LPLD Patients
Brief Title: Alipogene Tiparvovec for the Treatment of LPLD Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: uniQure, has decided not to renew the Marketing Authorization of Glybera in the EU. This decision is not related to any safety, efficacy or quality issue
Sponsor: UniQure Biopharma B.V. (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gly-CD-001
Record Dates: First submitted 2016-05-10; First posted 2016-09-19 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: LPL Deficiency
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Alipogene tiparvovec; Prednisolone; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- alipogene tiparvovec with IS (Other): Patients in the Immuno+ group will receive an immunosuppressant regimen to be initiated three days prior to alipogene tiparvovec administration. The regimen is to be continued for 12 weeks: Cyclosporins (3 mg/kg/day) and mycophenolate mofetil (2 x 1 g/day). Patients will receive IV bolus of 1mg/kg of methyl Prednisolone half an hour prior to IMP administration.
  Interventions: Drug: alipogene tiparvovec; Drug: Prednisolone; Drug: Cyclosporins; Drug: Mycophenolate mofetil
- alipogene tiparvovec without IS (Other): Patients in the Immuno- group will not receive an immunosuppressant regimen during 12 weeks. Patients will receive IV bolus of 1mg/kg of methyl Prednisolone half an hour prior to IMP administration.
  Interventions: Drug: alipogene tiparvovec; Drug: Prednisolone

INTERVENTIONS:
Drug: alipogene tiparvovec — A dose of 1x10(*12) gc/kg alipogene tiparvovec (Glybera) of body weight administered as a single set of intramuscular injections at multiple sites in multiple muscles of both upper legs and if necessary, the lower legs.
  Other Names: Glybera
Drug: Prednisolone — IV bolus methylprednisolone 1mg/kg half hour prior to administration
Drug: Cyclosporins — Immuno + group will receive cyclosporine (3 mg/kg/day) from three days prior to until 12 weeks following IMP administration
  Arms: alipogene tiparvovec with IS
Drug: Mycophenolate mofetil — Immuno + group will receive Mycophenolate mofetil (2x 1 g/day) from three days prior to until 12 weeks following IMP administration
  Arms: alipogene tiparvovec with IS

SUMMARY:
The aim of the study is to provide further confirmatory evidence of clinical benefit in LPLD patients treated with alipogene tiparvovec by assessing both the "clinical response" (as defined by a range of parameters), and "the metabolic response" (postprandial CM metabolism) in LPLD patients with and without an immunosuppressant regimen.

DETAILED DESCRIPTION:
This is a prospective, interventional, randomised, open-label, parallel group study evaluating the clinical response as well as the dynamics of postprandial chylomicron metabolism in patients treated with alipogene tiparvovec with and without immunosuppressants. The study will be conducted in 12 LPLD patients who will be randomised into the Immuno+ (cyclosporin and mycophenolate mofetil) or the Immuno- group.

ELIGIBILITY:
Main inclusion criteria are:

* Patients with a history of severe or multiple pancreatitis attacks despite dietary fat restriction.
* Genetically confirmed diagnosis of LPLD
* Post-heparin plasma LPL protein mass > 5% of normal
* LPL activity ≤20% of normal (in post- heparin plasma)
* Fasting plasma TG concentration >10 mmol/L.

Main exclusion criteria are:

* Females with a positive pregnancy test or who are breastfeeding, or on contraceptive use.
* Patients with a positive HIV, Hepatitis B, Hepatitis C or being positive for tuberculosis.
* Patients under treatment with antiplatelet or other anti-coagulants.
* Patient allergic to or having a condition that prohibits the use of immunosuppressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The Clinical Response of alipogene tiparvovec in LPLD patients | 2 years
  The overall clinical response of alipogene tiparvovec in LPLD patients will be assessed compared to baseline, by a combination of measurements, of which each gives relevant information to obtain enough and solid evidence in a small trial. Each of these outcome measures will be evaluated in combination with the results of other measures (to get an overall conclusion relating the clinical response). Descriptive methods will be used (so no formal statistical analyses will be performed), due to the specific nature and the small sample size of a rare disease trial.
The long term effect of alipogene tiparvovec on post prandial metabolism of chylomicrons (ppCM) in LPLD patients. | 2 years
  CM [3H]-activity will be assessed during ppCM testing pre- and post-dose, compared to baseline.

SECONDARY OUTCOMES:
The effect of alipogene tiparvovec on postprandial metabolism of chylomicrons (ppCM) in LPLD patients with and without immunosuppression treatment, at 14 weeks post-administration. | Baseline, 14 weeks
  CM [3H]-activity will be assessed during ppCM testing pre- and post-dose, compared to baseline.
Immuno response of alipogene tiparvovec by analysis of antibody formation | Baseline, 1 and 2 years post dose
  The immuno response of alipogene tiparvovec will be assessed by measuring the antibody formation compared to baseline.
Immuno response of alipogene tiparvovec by analysis of T-cell response | Baseline, 1 and 2 years post dose
  T-cell responses against alipogene tiparvovec will be assessed by measuring the T-cell response compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (2):
- Perelman School of Medicine at The University of Pennsylvania Translational Medicine & Human Genetics, Philadelphia, Pennsylvania, United States
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No